CLINICAL TRIAL: NCT03093376
Title: Neurally Targeted Interventions to Reduce Early Childhood Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan State University (Other); One Mind Institute (Unknown)
Responsible Party: Principal Investigator, Kate D. Fitzgerald, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00117593
Record Dates: First submitted 2017-01-30; First posted 2017-03-28 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Effortful Control; Preschool; ERN
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Child participants receive effortful control (EC) training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effortful Control Camp (Experimental): Children will participate in an interactive, child-friendly "camp" comprised of short, game-like exercises to teach inhibitory and attentional control, as well as visuospatial and working memory skills.
  Interventions: Behavioral: Effortful Control Camp

INTERVENTIONS:
Behavioral: Effortful Control Camp — An interactive, child-friendly "camp". Effortful control (EC) camp is comprised of short, game-like exercises taught by "camp counselors" to groups of approximately 4-6 children. In total, 12 different exercises that teach inhibitory and attentional control, as well as visuospatial and working memory skills, will be administered.
  Tasks will allow for "scaffolding" (Halperin et al, 2013), or incremental increases in difficulty of the games over time. EC camp will occur over 4 mornings from 9AM to 12PM, on two consecutive weekends.
  Other Names: EC Camp

SUMMARY:
Clinically significant anxiety affects up to 20% of preschool-aged children and often fails to respond to currently available treatments. Emerging science suggests that increasing brain capacity for "effortful control" (EC) may help anxious children to regulate emotion and behavior to improve outcomes. Thus, in the proposed study, children will be trained on EC tasks (including selective attention, response inhibition, etc.) to increase capacity for effortful control (EC) over fear behaviors. To determine whether EC training improves brain capacity to regulate fear, investigators will assess neurophysiological and behavioral indices of effortful control and fear reactivity before and after this training.

DETAILED DESCRIPTION:
8.4.21 Update: In late 2020, funding for a larger version of this study was received. Although originally intended to include randomization between active EC training and a waitlist control, this original pilot study was only able to collect data for the active EC training condition. The larger study (NCT04960813) recruits children to participate in a protocol with both the original EC training and an active play-based comparison group.

4.3.20 Update: Recruitment is ongoing. Enrollment and interactions are temporarily paused due to COVID-19. This is not a suspension of IRB approval.

This experiment examined child participants with clinical to subclinical anxiety to test the effects of a piloted effortful control (EC) training intervention. Up to 40 preschool age children (4-6.99 years) with clinical to subclinical anxiety symptoms were sought to complete a camp-like EC training (up to n=40). Before and after the intervention (time 1 and time 2, respectively), an EEG-based measure, the error-related negativity (ERN), was collected while children play a simple computer game. The ERN indexes neural mechanisms underlying EC. Other measures collected before and after the EC training included a blink reflex known as the fear potentiated startle (FPS); laboratory-assessed EC and fear behaviors; and, clinically assessed anxiety symptoms. Originally, the study was designed to include randomization between the EC training and a waitlist control; however, due to limited personnel and financial constraints, a decision was made to focus enrollment on the EC training.

The EC intervention or "EC camp" occurred over several sessions spread across 2 or more weeks. Times were chosen to maximize child focus and energy as well as convenience for families. EC camp was comprised of short, game-like exercises that teach effortful control skills (e.g., response inhibition, selective attention, set shifting skills).

As originally planned, primary analyses tested for group mean differences in ERN and FPS changes (i.e. from time 1 to time 2) among children assigned to EC training. Secondary analyses tested relationship of changes in neurophysiological targets with change in EC and Fear behaviors and change in anxiety severity.

This study was designed to examine the mechanistic plausibility of a precise, neuroscientifically-derived treatment for childhood anxiety, promoting developmental trajectories towards health and away from chronic illness.

ELIGIBILITY:
Inclusion Criteria:

* Children between 4.0 and 6.99 years
* Child has current anxiety symptoms
* Parent/caregiver is English-speaking.

Exclusion Criteria:

* Child cannot be currently taking medications that affect central nervous system functioning.
* No history of:

  * Head injury
  * Serious medical or neurological illness
  * Post-Traumatic Stress Disorder
  * Neurodevelopmental delay
  * Autism spectrum disorder (ASD)
  * Intellectual disability

Ages: 48 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Error Related Negativity (ERN) at Post-Intervention | approximately 10 weeks
  Error-related negativity (ERN) is assessed through the "Zoo task", a "Go/No-Go" paradigm assessing effortful control. Children view a series of animals on a computer screen and are asked to press a button when a new animal appears (Go trials), unless the animal is an orangutan (i.e., inhibit button response, No-Go trials). The task includes 8 blocks, each containing 30 unique animals (Go trials) and 10 orangutans (No-Go trials) in random order.
  Event related potentials (ERP; direct responses to stimuli measured using electroencephalography) will be examined from fronto-central recording sites time-locked to error and correct response. Differentiation between these trial types is the primary ERN measure, but ERN in error trials will also be considered, as well as ERPs in correct trials. The number of No-Go errors and response times (RTs) to Go trials will also be considered in analyses, as performance can affect ERN amplitude.
Change from Baseline Fear Potentiated Startle (FPS) at Post-Intervention | approximately 10 weeks
  Preschool participants watch age appropriate film clips (four fearful, four neutral, and four happy clips). White noise bursts are presented at varying time points to elicit the startle eyeblink response (FPS), recorded from two electrodes under the left eye.

SECONDARY OUTCOMES:
Change in Anxiety Symptoms | approximately 10 weeks
  Assessed using the Spence Anxiety Scale for Preschoolers (Spence, Rapee, McDonald, & Ingram, 2001). This 34-item parent-report scale provides an overall measure of child anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Kate D Fitzgerald, MD, Principal Investigator — University of Michigan; Maria Muzik, MD, Principal Investigator — University of Michigan; Kate Rosenblum, PhD, Principal Investigator — University of Michigan; Jason Moser, PhD, Principal Investigator — Michigan State University
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schroder HS, Ip KI, Hruschak JL, Horbatch F, Hall M, Liu Y, Mannella K, Muzik M, Rosenblum KL, Moser JS, Fitzgerald KD. Targeting cognitive control to reduce anxiety in very young children: A proof of concept study. Depress Anxiety. 2022 Aug;39(8-9):646-656. doi: 10.1002/da.23270. Epub 2022 Jun 16. PMID 35708131